CLINICAL TRIAL: NCT05406947
Title: Establishment and Clinical Application of Risk Classification Model Based on Molecular Typing of Medulloblastoma in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Neurosurgical Institute (Other); Beijing Children's Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Xuanwu Hospital, Beijing (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Tianyongji, Director, Beijing Tiantan Hospital
Other Study IDs: ChiCTR2200058760
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Medulloblastoma, Childhood
Keywords: Medulloblastoma; Glioma; Medulloblastoma, Childhood, Recurrent; Neuroepithelioma
MeSH Terms: conditions — Medulloblastoma; Glioma; Recurrence; Neuroectodermal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study, clinical samples (blood, cerebrospinal fluid, and tumor samples) are collected in the clinical working environment, and the samples are mainly from tumor tissues that must be removed during the operation and blood used for blood matching. The collection of cerebrospinal fluid is the remaining sample for clinical laboratory testing, and the damage to the patient is minimal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low risk group: Based on clinicopathological diagnosis and molecular pathological diagnosis, the children were classified into low risk groups, individualized radiotherapy and chemotherapy plan was made, and a perfect registration and follow-up system was established.
  Interventions: Other: Prospective observational study, no intervention
- Middle risk group: Based on clinicopathological diagnosis and molecular pathological diagnosis, the children were classified into middle risk groups, individualized radiotherapy and chemotherapy plan was made, and a perfect registration and follow-up system was established.
  Interventions: Other: Prospective observational study, no intervention
- High risk group: Based on clinicopathological diagnosis and molecular pathological diagnosis, the children were classified into high risk groups, individualized radiotherapy and chemotherapy plan was made, and a perfect registration and follow-up system was established.
  Interventions: Other: Prospective observational study, no intervention

INTERVENTIONS:
Other: Prospective observational study, no intervention — Prospective observational study, no intervention

SUMMARY:
The purpose of this study:(1) Development of a new risk classification model for childhood medulloblastoma. (2) Evaluation and improvement of existing individualized treatment protocols.

DETAILED DESCRIPTION:
Medulloblastoma (medulloblastoma, MB) is the most common intracranial malignant tumor in children, accounting for 20% of all central nervous system tumors in children, seriously affecting the quality of life and life span of children. Based on a retrospective analysis of previous MB cases in our center, we found that the clinical prognosis of previous MB patients in our center was worse than that in foreign countries, with an overall five-year survival rate of about 65%, and nearly 30% of the patients had tumor recurrence and metastasis within 2 years after the operation, and the prognosis was poor. We analyzed the possible reasons as follows: (1) the compliance to radiotherapy and chemotherapy in children with MB in our center was poor, and some of the patients only completed radiotherapy and had poor compliance with chemotherapy; (2) due to the lack of family doctor system, the tumor of the newly diagnosed patients was huge, which seriously affected the important brain function and clinical prognosis; (3) the patients were not followed up strictly and regularly after operation to monitor tumor recurrence, which led to poor treatment effect after recurrence.

(4) the unified treatment standard has not been formed yet, and the treatment mode for patients is complex.

As the largest neurosurgery and pediatric neurosurgery center in China, the center intends to prospectively establish a high-quality homogeneous MB observation cohort in children, make use of the center's case resources and biological sample processing advantages, and carry out accurate treatment research on children's MB through regular follow-up and systematic management of the clinical cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 0.5-18 years (except neonates).
* Pathologically confirmed medulloblastoma.
* Not having received any other relevant treatment before surgery.
* Completion of enhanced MRI of the head and spinal cord.
* Availability of tumor samples and determination of molecular typing.
* Postoperative KPS score ≥ 70.
* Voluntary enrollment in the group and the ability to receive long-term follow-up.
* The patient or the patient's family voluntarily signed the informed consent form.

Exclusion Criteria:

* Patients who have recently received other drugs or radiation therapy.
* Patients suffering from acute or chronic infectious diseases
* Patients suffering from neurological or psychiatric diseases or mental disorders that cannot be easily controlled, or poor compliance.
* Patients who cannot receive enhanced MRI scans.
* Other conditions that the investigator believes make the patient unfit to participate in this trial.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 350 medulloblastoma patients aged 0.5-18 years (except newborns)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular typing | 2022-2030
  Medulloblastoma can be classified into four molecular types: WNT, SHH, G3 and G4.
Overall survival | 2022-2030
  the time from operation to death
Progression free survival | 2022-2030
  The time from operation to disease progression
Quality of life scale | 2022-2030
  A scale for evaluating the quality of life of patients after operation
Adjunctive treatment | 2022-2030
  Patients receive postoperative radiotherapy or chemotherapy

SECONDARY OUTCOMES:
Age at diagnosis | 2022-2030
BMI | 2022-2030
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Yongji Tian, MD, Principal Investigator — Beijing TianTanHospital, China Capital Medical University; FU ZHAO, MD, Principal Investigator — Beijing Neurosurgical Institute

IPD SHARING:
Plan to Share IPD: Undecided